CLINICAL TRIAL: NCT06576856
Title: Use of Salivary Markers to Heralding the Onset of Periodontal Disorders
Brief Title: Salivary Markers in Periodontal Disorders
Status: Completed | Type: Observational
Sponsor: Midwestern University (Other)
Responsible Party: Sponsor
Other Study IDs: 20082
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Periodontal Disease, Staging, Salivary Markers, Diagnosis
MeSH Terms: conditions — Periodontal Diseases; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Salivary samples without DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Perio-Healthy: Individuals included in this cohort, other than meet the eligibility criteria, should present no clinical sign of periodontal disease. We anticipate to find from a very small number to none participants at this cohort. No intervention are anticipated.
  Interventions: Other: This is an observational study, no intervention is anticipated.
- Periodontitis Stage I: Individuals included in this cohort, other than meet the eligibility criteria, should present clinical sign of periodontal defined as Stage I according to the American Academy of Periodontology. We anticipate low to moderate number of participants in this cohort. No interventions are anticipated.
  Interventions: Other: This is an observational study, no intervention is anticipated.
- Periodontitis Stage II: Individuals included in this cohort, other than meet the eligibility criteria, should present clinical sign of periodontal defined as Stage II according to the American Academy of Periodontology. We anticipate a moderate number of participants in this cohort. No interventions are anticipated.
  Interventions: Other: This is an observational study, no intervention is anticipated.
- Periodontitis Stage III: Individuals included in this cohort, other than meet the eligibility criteria, should present clinical sign of periodontal defined as Stage III according to the American Academy of Periodontology. We anticipate moderate to high number of participants in this cohort. No interventions are anticipated.
  Interventions: Other: This is an observational study, no intervention is anticipated.
- Periodontitis Stage IV: Individuals included in this cohort, other than meet the eligibility criteria, should present clinical sign of periodontal defined as Stage IV according to the American Academy of Periodontology. We anticipate low to moderate number of participants in this cohort. No interventions are anticipated.
  Interventions: Other: This is an observational study, no intervention is anticipated.

INTERVENTIONS:
Other: This is an observational study, no intervention is anticipated. — There is no intervention. This is an observational study.

SUMMARY:
The swelling of the gum, or periodontitis, is the leading cause for tooth loss, and currently affects up to 65 million adults only in the United States. One of the reasons for the widespread of periodontitis is because currently there are no definitive methods to detect the onset of gum disease. This lack of foresight impedes medical professionals to enact any preventive measures before the disease already manifests itself.

We wish to expand our understanding towards the development of periodontitis by studying the expression and activity of salivary markers that have been associated with advanced stages of the disease, wherein the supporting tissues of tooth (periodontium) are already irreversibly destroyed. We hypothesize that a progressive shift in the expression of such salivary markers can indicate a change or evolution of periodontitis staging.

In specific, we seek to establish a quantifiable relationship among levels of salivary proteases called MMPs, level of metal ions in different stages varying from health to periodontitis. The overall goal of this proposal is to enhance the predictability of periodontitis, as we are currently unable to diagnose the disease until the manifestation of its clinical signs and symptoms.

DETAILED DESCRIPTION:
There is an urgent need for an efficient system to diagnose periodontal disease in its early stages. A recent investigation on the prevalence of periodontitis in adults living in the USA revealed that almost 50% of the assayed individuals had periodontal disease. Research on the economic burden of oral diseases estimated that productivity losses due to severe periodontitis and, consequently, due to tooth loss in North America (US and Canada) amounted US$ 116 billion yearly. This pervasiveness of periodontitis can be attributed to the conventional method of diagnosis, which is entirely based upon recognizing observable signs - an assessment of the disease's history.

A crucial restraint of these observable parameters is that they do not detect present disease activity and, therefore, cannot provide a real-time evaluation of the disease status. The lack of evidence-based knowledge regarding periodontal diseases activity and level of progression may ultimately lead to unintentional clinical mismanagement [6]. Accordingly, there is an unmet requisite for easy and readily available methods to herald the periodontium health condition prior to the manifestation of disease clinical signs [7].

Periodontal diseases are identified as being resultant from an inflammatory, host-mediated response, associated with dysbiotic plaque biofilms. Within the inflammatory host response of periodontal diseases there is a group of enzymes that are key, the matrix metalloproteinases (MMP). The abundance of MMPs, more specifically MMP-8, in saliva of individuals with severe periodontitis has shown to be high. In physiological conditions, the activity of MMPs is tightly controlled by changes in the balance between their expression and the expression of their major tissue endogenous inhibitors, called TIMPs. In addition, the catalytic competence of MMPs is highly dependent on the concentration of specific metal ions, zinc and calcium, which justifies the use of the prefix "metal" to classify and group this proteinase superfamily. As MMP-inhibitory medication has been shown to reduce the levels of MMPs in oral fluids, we hypothesize that collection of oral fluid samples (i.e., saliva and/or gingival crevicular fluid) from individuals appertaining to different stages of periodontal diseases can identify a shift in the balance between MMPs and their tissue-regulatory factors.

The overall objective of this proposal is to contribute to enhance the predictability of periodontitis and identify a method to heralding its onset. We hypothesize that the levels of salivary MMPs and other factors modulating these enzymes activity relate with different clinical stages of periodontal disease. The questions this research will address are: Do the level of MMPs vary as a function of periodontium health state? Is there a quantifiable relationship between salivary MMPs and other markers, such as MMP-Tissue Inhibitors (TIMPs) and metal ions, in the context of periodontitis?

Thus, the specific aims of this purposed study are:

* To measure the levels of MMPs and MMPs' tissue-regulatory factors (TIMPs and metal ions) in oral fluids of adults displaying different clinical status of periodontium integrity, from health (stage 0) to severe periodontitis (stage IV).
* To determine the relationship of periodontitis clinical staging and levels of salivary MMPs and MMPs regulatory factors.

ELIGIBILITY:
Inclusion Criteria:

* (1) 40 years of age or older with a healthy medical history and not meeting any of the exclusion criteria;
* (2) requiring definitive periodontal treatment/routine care; and
* (3) retaining a minimum of 20 teeth and without active carious lesions

Exclusion Criteria:

* 1) with systemic illness affecting their immune system (i.e. diabetes, rheumatoid arthritis, etc);
* (2) currently on chronic anti-inflammatory medications (i.e. steroids, TNFα-inhibitors, etc); and
* (3) previously underwent active periodontal therapy within the past 2 years;
* (4) who cannot read or speak English.

Ages: 30 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The literature does not display a consistent number of estimate participants for reliable assessment of salivary markers; with correlate studies reporting to have included from 100 to 1000 participants. We aim to invite up to 200 subjects to participate in this research. Subjects will be allocated into four categories following the four stages of periodontitis from AAP classification, plus a fifth category as periodontal health individuals for control group. The results of this cohort will be analyzed to detect an effect size of 0.5 at the 0.05 significance level.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-11-06 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Matrix Metalloproteases (MMPs) Salivary Levels | October 2024
  Levels of MMPs assessed by different immuno-assays.
Levels of Metal Ions | October 2024
  Levels of metal ions assessed by Inductively Coupled Plasma Dynamic Reaction Cell Mass Spectrometer

SECONDARY OUTCOMES:
Potential Correlation of MMPs, Metal Ions and Peridontitis Staging | October 2024
  The relationship between salivary MMPs and identified metal ions for all cohorts (periodontally healthy and periodontitis-affected individuals) will be determined by multiple regression analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Rocha de Oliveira Carrilho, DDS, PhD, Principal Investigator — Midwestern University
Locations (1):
- Midwestern Univerity, Downers Grove, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not make available to other researchers.

REFERENCES:
- [Background] Butler GS, Overall CM. Matrix metalloproteinase processing of signaling molecules to regulate inflammation. Periodontol 2000. 2013 Oct;63(1):123-48. doi: 10.1111/prd.12035. PMID 23931058
- [Background] de Morais EF, Pinheiro JC, Leite RB, Santos PPA, Barboza CAG, Freitas RA. Matrix metalloproteinase-8 levels in periodontal disease patients: A systematic review. J Periodontal Res. 2018 Apr;53(2):156-163. doi: 10.1111/jre.12495. Epub 2017 Sep 12. PMID 28898418
- [Background] Sorsa T, Gursoy UK, Nwhator S, Hernandez M, Tervahartiala T, Leppilahti J, Gursoy M, Kononen E, Emingil G, Pussinen PJ, Mantyla P. Analysis of matrix metalloproteinases, especially MMP-8, in gingival creviclular fluid, mouthrinse and saliva for monitoring periodontal diseases. Periodontol 2000. 2016 Feb;70(1):142-63. doi: 10.1111/prd.12101. PMID 26662488
- [Background] Sorsa T, Tjaderhane L, Salo T. Matrix metalloproteinases (MMPs) in oral diseases. Oral Dis. 2004 Nov;10(6):311-8. doi: 10.1111/j.1601-0825.2004.01038.x. PMID 15533204
- [Background] Schwarz F, Derks J, Monje A, Wang HL. Peri-implantitis. J Periodontol. 2018 Jun;89 Suppl 1:S267-S290. doi: 10.1002/JPER.16-0350. PMID 29926957
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S173-S182. doi: 10.1002/JPER.17-0721. PMID 29926951
- [Background] Giannobile WV, Beikler T, Kinney JS, Ramseier CA, Morelli T, Wong DT. Saliva as a diagnostic tool for periodontal disease: current state and future directions. Periodontol 2000. 2009;50:52-64. doi: 10.1111/j.1600-0757.2008.00288.x. No abstract available. PMID 19388953
- [Background] Slots J. Periodontology: past, present, perspectives. Periodontol 2000. 2013 Jun;62(1):7-19. doi: 10.1111/prd.12011. PMID 23574461
- [Background] Kwok V, Caton JG, Polson AM, Hunter PG. Application of evidence-based dentistry: from research to clinical periodontal practice. Periodontol 2000. 2012 Jun;59(1):61-74. doi: 10.1111/j.1600-0757.2011.00437.x. PMID 22507060
- [Background] Lang NP, Tonetti MS. Periodontal diagnosis in treated periodontitis. Why, when and how to use clinical parameters. J Clin Periodontol. 1996 Mar;23(3 Pt 2):240-50. doi: 10.1111/j.1600-051x.1996.tb02083.x. PMID 8707984
- [Background] Ji S, Choi Y. Point-of-care diagnosis of periodontitis using saliva: technically feasible but still a challenge. Front Cell Infect Microbiol. 2015 Sep 3;5:65. doi: 10.3389/fcimb.2015.00065. eCollection 2015. PMID 26389079
- [Background] Listl S, Galloway J, Mossey PA, Marcenes W. Global Economic Impact of Dental Diseases. J Dent Res. 2015 Oct;94(10):1355-61. doi: 10.1177/0022034515602879. Epub 2015 Aug 28. PMID 26318590
- [Background] Eke PI, Dye BA, Wei L, Slade GD, Thornton-Evans GO, Borgnakke WS, Taylor GW, Page RC, Beck JD, Genco RJ. Update on Prevalence of Periodontitis in Adults in the United States: NHANES 2009 to 2012. J Periodontol. 2015 May;86(5):611-22. doi: 10.1902/jop.2015.140520. Epub 2015 Feb 17. PMID 25688694
- See also: . Many matrix metalloproteinase substrates modulate inflammation and hence, by processing these proteins, matrix metalloproteinases can orchestrate the inflammatory response. — https://pubmed.ncbi.nlm.nih.gov/23931058/